CLINICAL TRIAL: NCT00286169
Title: Randomized Phase III Trial of Amrubicin Versus Carboplatin Plus Etoposide in Elderly Patients With Extensive-disease Small-cell Lung Cancer
Brief Title: Amrubicin Study for Elderly Patients With Extensive-disease Small-cell Lung Cancer (ED-SCLC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D0702002; JapicCTI-060203
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Small-cell Lung Cancer
Keywords: Extensive-disease small-cell lung cancer (ED-SCLC)
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — amrubicin

INTERVENTIONS:
Drug: Amrubicin Hydrochloride

SUMMARY:
The purpose of this study is to compare the efficacy and toxicity of amrubicin with carboplatin plus etoposide in elderly patients with extensive-disease small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Extensive-disease small-cell lung cancer
* Aged 70 years or older
* Performance status of 0-2
* No prior chemotherapy

Exclusion Criteria:

* Prior therapy for primary lesion
* Pneumonitis and/or pulmonary fibrosis
* Active concomitant malignancy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2006-04

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Time to progression
Objective tumor response
Quality of Life (QOL: EuroQOL, FACT-L-LCS)
Frequency and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Drug Development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (8):
- Japan (8):
  - Chugoku Region Site, Chugoku
  - Chubu Region Site, Chūbu
  - Hokkaido Region Site, Hokkaido
  - Kanto Region Site, Kanto
  - Kinki Region Site, Kinki
  - Kyushu Region Site, Kyushu
  - Shikoku Region Site, Shikoku
  - Tohoku Region Site, Tōhoku